CLINICAL TRIAL: NCT04010240
Title: A Study to Determine the Incidence of NTRK Fusions in Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors With NTRK Fusions and Related Treatment Outcomes.
Brief Title: A Retrospective Study to Determine the Incidence of NTRK Fusions. NTRK Study
Acronym: NTRK
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: IB2015-NTRK; MR 0112040319 (Other: Insitut National des Données de Santé (INDS))
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Solid Tumors
Keywords: Solid tumor; Metastatic; NTRK
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Parrafin embedded tumor material
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors
  Interventions: Other: No intervention (this is a retrospective cohort study)

INTERVENTIONS:
Other: No intervention (this is a retrospective cohort study) — No intervention (this is a retrospective cohort study) aimed at describing tumour samples. No treatment/intervention is being tested.

SUMMARY:
This retrospective study has a primary objective to estimate the incidence of NTRK gene fusion depending on the histological diagnosis.

DETAILED DESCRIPTION:
This retrospective study has a primary objective to estimate the incidence of NTRK gene fusion depending on the histological diagnosis. The tropomyosin receptor kinase (Trk) receptor family comprises 3 transmembrane proteins referred to as Trk A, B and C (TrkA, TrkB and TrkC) receptors that are encoded by the NTRK1, NTRK2 and NTRK3 genes, respectively. These receptor tyrosine kinases are expressed in human neuronal tissue and play an essential role in the physiology of development and function of the nervous system through activation by neurotrophins. Gene fusions involving NTRK genes lead to transcription of chimeric Trk proteins with constitutively activated or overexpressed kinase function conferring oncogenic potential. These genetic abnormalities have recently emerged as targets for cancer therapy, because novel compounds have been developed that are selective inhibitors of the constitutively active rearranged proteins. Developments in this field are being aided by next generation sequencing methods as tools for unbiased gene fusions discovery. However, the incidence of NTRK aberrations in solid tumors is unknown as well as the natural history of NTRK-rearranged tumors This study will provide better knowledge of NTRK gene fusion incidence to allow recommendations for pathological diagnosis.

Subjects who are tested positive by Immunohistochemistry (IHC : Pan-Trk IHC testing with mAb EPR17341) will be the subject of molecular assays such as next-generation sequencing (Archer Dx fusion assay) of tumor material [parrafin embedded material]), so that tumor harboring NTRK1, NTRK2 or NTRK3 gene fusions, is identified properly.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 1 month.
* Subject has/had a histologically or cytologically confirmed diagnosis of solid tumor including but not exclusively: soft tissue sarcoma, BRAF wild type melanoma, KRAS wild-type colorectal cancer, central nervous system, EGFR-wild type non-small cell lung cancer.
* Subject has locally advanced/unresectable or metastatic disease.
* Subject has received at least one systemic anti-cancer therapy for locally advanced/unresectable or metastatic disease for which there is available outcome information in terms of PFS, or the latter can be estimated based on the subject's records.
* Subject has tumor material available for immunoscreening (IHC for NTRK gene fusions).
* Written and voluntary informed consent understood, signed and dated, or a waiver of consent is granted according to French régulations.

Exclusion Criteria:

• Subjects who have not yet received or completed at least one systemic anti-cancer therapy for locally advanced/unresectable or metastatic cancer.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort will included both adult and pediatric patients with metastatic solid tumors, who have received at least one systemic anti-cancer therapy for advanced disease and for which there is available both outcome information and tumor material.
Sampling Method: Non-Probability Sample
Enrollment: 3820 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ITALIANO, MD, PhD, Principal Investigator — a.italiano@bordeaux.unicancer.fr
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Retrospective Cohort: For eligible subject, tumor material will be tested by immunohistochemistry (Pan-Trk ICH testing with mAb EPR17341).
  Retrospective cohort: Tumor material tested positive will be analyzed by next-generation sequencing to identify NTRK1, NTRK2 or NTRK3 gene fusions.
Period: Overall Study
Arm/Group | Retrospective Cohort
Started | 3820
Completed | 1521
Not Completed | 2299
Not completed — IHC not performed | 2299

BASELINE CHARACTERISTICS:
Population: Age and sex were not collected.
Groups:
- Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors: Tumor material was tested by immunohistochemistry (Pan-Trk ICH testing with mAb EPR17341). Tumor material tested positive were analyzed by next-generation sequencing to identify NTRK1, NTRK2 or NTRK3 gene fusions.
Arm/Group | Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors
Number analyzed (Participants) | 3820
Age, Categorical [Count of Participants; unit: Participants] — Population: Age was not collected
Sex: Female, Male [Count of Participants; unit: Participants] — Sex was not collected Population: Sex was not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 3820

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With NRTK Fusions Among Participants Analyzed by NGS (Next-generation Sequencing).
Description: A participant with NRTK fusion is defined as a participant with a tumor harboring NTRK1, NTRK2 or NTRK3 gene fusions, based on NGS (Next-generation sequencing methods).
  NGS (Next-generation sequencing methods) method: DNA and RNA were extracted from tumor tissue according to standard procedures. All samples had their RNA analyzed with Archer or full RNA sequencing to assess specific novel NTRK1, 2, and 3 rearrangements for the production of NTRK fusion transcripts. Alternatively, DNA was analyzed by using an hybrid-capture based NGS assay as previously described.
Time Frame: at baseline (i.e. at the time of tumor removal)
Population: Subjects with locally advanced/unresectable or metastatic solid tumors and for whom NGS (new generation sequencing) was performed
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors and NGS Performed.: NGS / Next-generation sequencing methods :
  DNA and RNA were extracted from tumor tissue according to standard procedures. All samples had their RNA analyzed with Archer or full RNA sequencing to assess specific novel NTRK1, 2, and 3 rearrangements for the production of NTRK fusion transcripts. Alternatively, DNA was analyzed by using an hybrid-capture based NGS assay.
Arm/Group | Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors and NGS Performed.
Number analyzed (Participants) | 2378
Participants | 11

2. Secondary Outcome: Count of Participants With NRTK Fusions Among Participants With With Positive Immunohistochemistry (IHC)
Description: A participant with NRTK fusion is defined as a participant with a tumor harboring NTRK1, NTRK2 or NTRK3 gene fusions, based on Immunohistochemistry (IHC).
  Immunohistochemistry (IHC) mehtod : Pan-TRK: rabbit monoclonal antibody, clone C17F1, Cell signaling dilution 1/50°. Automate Benchmark: ULTRA Ventana, CC1 64', incubation 52', revelation kit Optiview
Time Frame: at baseline (i.e. at the time of tumor removal)
Population: Participants with positive IHC results
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors: Subjects with locally advanced/unresectable or metastatic solid tumors anf for whom NGS (new generation sequencing) and IHC were performed
Arm/Group | Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors
Number analyzed (Participants) | 79
Participants | 1

3. Other Pre Specified Outcome: Progression-free Survival (PFS) in Patients With NRTK Gene Fusion.
Description: PFS is calculated using Kaplan-Meier method, in the population of patients with positive IHC results.
Time Frame: Two years after tumor removal
Population: Only one patient had positive IHC results and had a gene NRTK fusion.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors
Number analyzed (Participants) | 1
years | NA — insufficient number of participants with events : There was only 1 patient with positive IHC results and had a gene NRTK fusion.

ADVERSE EVENTS:
Time Frame: Retrospective NGS analysis. AE were not collected
Description: AE were not collected
Groups:
- Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors: Retrospective cohort: For eligible subject, tumor material will be tested by immunohistochemistry (Pan-Trk ICH testing with mAb EPR17341). Tumor material tested positive will be analyzed by next-generation sequencing to identify NTRK1, NTRK2 or NTRK3 gene fusions.
Arm/Group | Subjects With Locally Advanced/Unresectable or Metastatic Solid Tumors
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT04010240/Prot_SAP_000.pdf